CLINICAL TRIAL: NCT05548907
Title: Sleep Restriction Treatment for Insomnia: a Randomized Controlled Trial
Brief Title: Sleep Restriction Treatment for Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Jaap Lancee, Assistant Professor, University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-CP-15342
Record Dates: First submitted 2022-09-06; First posted 2022-09-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Insomnia
Keywords: insomnia; behavioral treatment; randomized controlled trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial where participants are allocated to either a sleep restriction treatment condition or a sleep monitoring control condition. All participants keep a daily sleep diary and fill out weekly questionnaires
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep restriction treatment (Experimental): In this condition participants receive a behavioral sleep restriction intervention for six weeks
  Interventions: Behavioral: sleep restriction treatment
- Sleep monitoring (Placebo Comparator): In this control condition people fill out a sleep diary for six weeks
  Interventions: Behavioral: sleep diary monitoring

INTERVENTIONS:
Behavioral: sleep restriction treatment — Treatment consists of sleep restriction treatment for insomnia. In this treatment, participants limit their bedtimes to the time they actually sleep. If they sleep most of the time in bed again then bedtimes are slowly built up again. This treatment technique has already been studied in several trials and found to be effective.
  Mode of delivery is an online booklet, online exercises and weekly telephone support
  Arms: Sleep restriction treatment
Behavioral: sleep diary monitoring — As an active control condition people monitor their sleep with a sleep diary (also included in the sleep restriction intervention)
  Arms: Sleep monitoring

SUMMARY:
With a prevalence of about 10% chronic insomnia is a common problem. The standard treatment for insomnia is cognitive behavioral therapy. According to many, the core element within this treatment is sleep restriction. This element has been examined separately in a couple of studies and also appears to be effective in isolation. In the current study the aim is to get more information about the effectiveness of this core element of the treatment. For this reason, a randomized study is conducted to compare sleep restriction with a diary control condition.

The second aim in this study is to determine mechanisms behind treatments. Network intervention analysis will be used to determine which specific symptoms are associated with therapy success. This is the reason that throughout the study weekly and daily measures will be conducted.

The expectations are that:

* Participants in the sleep restriction condition will improve more on insomnia complaints than the sleep diary control condition (primary outcome)
* Participants in the sleep restriction condition will improve more on sleep diary outcomes and other secondary outcomes compared to the sleep diary control condition (secondary outcome)

ELIGIBILITY:
Inclusion Criteria:

* Insomnia Severity Index Score ≥ 10
* 18 years or older
* Self reported insomnia complaints: being awake ≥30 minutes per night, ≥3 nights per week, ≥ 3 months
* Daytime problems related to sleep complaints
* Sleep efficiency < 85%
* Dutch speaking

Exclusion Criteria:

* (1) No acces to internet
* (2) Pregnant or breastfeeding
* (3) working in night shifts
* (4) currently in psychological treatment (started < 6 months) or on wait-list for treatment
* (5) cognitive behavioral treatment for insomnia in last 12 months
* (6) concrete suicidal ideation
* (7) schizophrenic or psychotic disorder
* (8) high level of depressive complaints (BDI-II > 28)
* (9) Instable medication use (medication should not be tampered in last 6 weeks) incidental sleep-medication use is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-11-11 (Actual); Study Completion 2023-11-11 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | Change from baseline to six weeks post-randomization
  The Insomnia Severity Index is a seven item-scale scored on a five-point Likert scale (Bastien et al. 2001). The total score ranges from 0 to 28. Higher scores indicate more insomnia.

SECONDARY OUTCOMES:
Sleep diary: sleep onset latency | Change from baseline to six-weeks post-randomization
  Sleep onset latency is assessed with the Carney (2012) consensus sleep diary. This is measured in minutes (higher scores indicating longer sleep onset latency).
Sleep diary: sleep onset latency | Change from baseline to six-month follow-up (intervention only)
  Sleep onset latency is assessed with the Carney (2012) consensus sleep diary. This is measured in minutes (higher scores indicating longer sleep onset latency).
Sleep diary: wake after sleep onset | Change from baseline to six-weeks post-randomization
  Wake after sleep onset is assessed with the Carney (2012) consensus sleep diary. This is measured in minutes (higher scores indicating longer wake after sleep onset).
Sleep diary: wake after sleep onset | Change from baseline to six-month follow-up (intervention only)
  Wake after sleep onset is assessed with the Carney (2012) consensus sleep diary. This is measured in minutes (higher scores indicating longer wake after sleep onset )
Sleep diary: terminal wakefulness | Change from baseline to six-weeks post-randomization
  Terminal wakefulness is assessed with the Carney (2012) consensus sleep diary. This is measured in minutes (higher scores indicating longer terminal wakefulness).
Sleep diary: terminal wakefulness | Change from baseline to six-month follow-up (intervention only)
  Terminal wakefulness is assessed with the Carney (2012) consensus sleep diary. This is measured in minutes (higher scores indicating longer terminal wakefulness).
Sleep diary: sleep efficiency | Change from baseline to six-weeks post-randomization
  Sleep efficiency is assessed with the Carney (2012) consensus sleep diary. This is measured in percentage (higher scores indicating better sleep efficiency).
Sleep diary: sleep efficiency | Change from baseline to six-month follow-up (intervention only)
  Sleep efficiency is assessed with the Carney (2012) consensus sleep diary. This is measured in percentage (higher scores indicating better sleep efficiency).
Sleep diary: total sleep time | Change from baseline to six-weeks post-randomization
  Total sleep time is assessed with the Carney (2012) consensus sleep diary. This is measured in minutes (higher scores indicating longer total sleep time).
Sleep diary: total sleep time | Change from baseline to six-month follow-up (intervention only)
  Total sleep time is assessed with the Carney (2012) consensus sleep diary. This is measured in minutes (higher scores indicating longer total sleep time).
Sleep diary: time in bed | Change from baseline to six-weeks post-randomization
  Time in bed is assessed with the Carney (2012) consensus sleep diary. This is measured in minutes (higher scores indicating longer time in bed).
Sleep diary: time in bed | Change from baseline to six-month follow-up (intervention only)
  Time in bed is assessed with the Carney (2012) consensus sleep diary. This is measured in minutes (higher scores indicating longer time in bed).
Cognitive arousal | Change from baseline to six weeks post randomization
  cognitive arousal is measured daily with a visual analogue scale
Somatic arousal | Change from baseline to six weeks post randomization
  Somatic arousal is measured daily with a visual analogue scale
Current sleepiness | Change from baseline to six weeks post randomization
  Sleepiness is measured daily with a visual analogue scale
Insomnia Severity | Change from baseline to six-month follow-up (intervention only)
  The Insomnia Severity Index is a seven item-scale scored on a five-point Likert scale (Bastien et al. 2001). The total score ranges from 0 to 28. Higher scores indicate more insomnia.
Sleep safety | Change from baseline to six weeks post-randomization
  Sleep safety behaviors are measured with the Dutch translation of the 32-item Sleep-Related Behaviors Questionnaire-SRBQ (Ree & Harvey, 2004). The total score ranges from 0 (no safety behaviors) to 128 (severe safety behaviors).
Sleep safety | Change from baseline to six-month follow-up (intervention only)
  Sleep safety behaviors are measured with the Dutch translation of the 32-item Sleep-Related Behaviors Questionnaire-SRBQ (Ree & Harvey, 2004). The total score ranges from 0 (no safety behaviors) to 128 (severe safety behaviors).
Epworth Sleepiness Scale | Change from baseline to six weeks post-randomization
  To assess daytime sleepiness the Epworth Sleepiness Scale (ESS) is used. The ESS consists of 8-items on a 4-point Likert scale (range 0-24) with higher scores indicating more sleepiness.
Epworth Sleepiness Scale | Change from baseline to six-month follow-up (intervention only)
  To assess daytime sleepiness the Epworth Sleepiness Scale (ESS) is used. The ESS consists of 8-items on a 4-point Likert scale (range 0-24) with higher scores indicating more sleepiness.
Pre-sleep arousal | Change from baseline to six weeks post-randomization
  Sleep-related arousal was measured with the Pre-sleep Arousal Scale (PSAS) (Nicassio et al. 1985). The PSAS consists of 16 items that range from 1 ('not at all') to 5 ('extremely'), higher scores indicating more arousal (range 16-80).
Pre-sleep arousal | Change from baseline to six-month follow-up (intervention only)
  Sleep-related arousal was measured with the Pre-sleep Arousal Scale (PSAS) (Nicassio et al. 1985). The PSAS consists of 16 items that range from 1 ('not at all') to 5 ('extremely'), higher scores indicating more arousal (range 16-80).
Sleep-bed association | Change from baseline to six weeks post-randomization
  Sleep-bed association is measured with a newly constructed scale of 5 items on a 7-point Likert scale (0-6). Higher scores indicating a stronger sleep-bed association (range 0-30)
Sleep-bed association | Change from baseline to six-month follow-up (intervention only)
  Sleep-bed association is measured with a newly constructed scale of 5 items on a 7-point Likert scale (0-6). Higher scores indicating a stronger sleep-bed association (range 0-30)
Dysfunctional beliefs | Change from baseline to six weeks post-randomization
  Dysfunctional beliefs about sleep are measured using the 16-item Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS-16) (Morin et al. 2017). Items are scored on an 11-point Likert scale (0-10). Higher scores indicating more dysfunctional beliefs (range 0-160).
Dysfunctional beliefs | Change from baseline to six-month follow-up (intervention only)
  Dysfunctional beliefs about sleep are measured using the 16-item Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS-16) (Morin et al. 2017). Items are scored on an 11-point Likert scale (0-10). Higher scores indicating more dysfunctional beliefs (range 0-160).
Depression | Change from baseline to six weeks post-randomization
  Depression is measured with the Dutch version of a nine-item depression scale, the Patient Health Questionnaire-9 (PHQ-9; range 0-27, Cronbach's α = 0.94; Spitzer et al., 1999). Higher scores indicating more depression.
Depression | Change from baseline to six-month follow-up (intervention only)
  Depression is measured with the Dutch version of a nine-item depression scale, the Patient Health Questionnaire-9 (PHQ-9; range 0-27, Cronbach's α = 0.94; Spitzer et al., 1999). Higher scores indicating more depression.
Anxiety | Change from baseline to six weeks post-randomization
  Anxiety is measured with the Anxiety section of the Hospital Anxiety and Depression Scale (HADS-A; Cronbach's α = 0.84, seven items on a four-point Likert scale, scores ranging 0-21; Spinhoven et al., 1997). Higher scores indicating more anxiety.
Anxiety | Change from baseline to six-month follow-up (intervention only)
  Anxiety is measured with the Anxiety section of the Hospital Anxiety and Depression Scale (HADS-A; Cronbach's α = 0.84, seven items on a four-point Likert scale, scores ranging 0-21; Spinhoven et al., 1997). Higher scores indicating more anxiety.
Acceptance | Change from baseline to six weeks post-randomization
  Acceptance is measured with 10-items of the 'flexibiliteits index test'. Items are scored on a 7-point Likert scale (0-6) and higher scores indicate more acceptance (range 0-60).
Acceptance | Change from baseline to six-month follow-up (intervention only)
  Acceptance is measured with 10-items of the 'flexibiliteits index test'. Items are scored on a 7-point Likert scale (0-6) and higher scores indicate more acceptance (range 0-60).
Adverse events | Six-weeks post-randomization
  Participants asked to report adverse events ("Did anything unpleasant happen to you that was related to your sleep or participation in the trial?"
Treatment quality | Six-weeks post-randomization
  Treatment quality is rated with a single question 'how do you rate the treatment'. This is rated on an 11-point Likert scale (0-10) with higher scores indicating more satisfaction (intervention only)
Rating coach | Six-weeks post-randomization
  Coaches are rated with a single question 'how satisfied were you with your coach during the treatment'. This is rated on an 11-point Likert scale (0-10) with higher scores indicating more satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Lancee, PhD, Principal Investigator — University of Amsterdam
Locations (1):
- University of Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data will be available upon requests

REFERENCES:
- [Derived] Looman MI, Blanken TF, Schoenmakers TM, Reesen JE, Effting M, Linnebank FE, van Straten A, Kamphuis JH, Lancee J. Telephone-Guided Sleep Restriction for Insomnia: A Randomized Sleep Diary-Controlled Trial. Psychother Psychosom. 2025;94(3):147-161. doi: 10.1159/000545138. Epub 2025 Mar 21. PMID 40122034